CLINICAL TRIAL: NCT02261727
Title: The Effect of Low-dose Corticosteroids and Theophylline on the Risk of Acute Exacerbations of COPD: the TASCS Randomised Clinical Trial
Brief Title: Theophylline and Steroids in Chronic Obstructive Pulmonary Disease (COPD) Study
Acronym: TASCS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TGI-Resp-01; 1033117 (Other Grant/Funding Number: National Health and Medical Research Council, Australia)
Record Dates: First submitted 2014-05-07; First posted 2014-10-10 (Estimated); Results first posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Theophylline; Oral corticosteroids; COPD exacerbations
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Theophylline; Prednisone; Cortisone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo theophylline, one tablet twice daily, and Placebo prednisone, one tablet once daily
  Interventions: Drug: Placebo (for prednisone); Drug: Placebo (for Theophylline)
- Low-dose theophylline arm (Active Comparator): Theophylline 100 mg twice daily
  Interventions: Drug: Theophylline; Drug: Placebo (for prednisone)
- Theophylline and Prednisone arm (Active Comparator): Theophylline 100 mg twice daily plus prednisone 5 mg once daily
  Interventions: Drug: Theophylline; Drug: Prednisone

INTERVENTIONS:
Drug: Theophylline — Theophylline is an oral methylxanthine which relaxes smooth muscle through its action as a phosphodiesterase inhibitor
  Other Names: Theophylline (100 mg twice a day)
  Arms: Low-dose theophylline arm; Theophylline and Prednisone arm
Drug: Prednisone — Prednisone is an oral glucocorticosteroid which has anti-inflammatory properties
  Other Names: Prednisone (5mg once daily); cortisone
  Arms: Theophylline and Prednisone arm
Drug: Placebo (for prednisone) — * Arm 1 : Theophylline Placebo 1 tab twice daily and Prednisone placebo 1 tab once daily
  * Arm 2 : Theophylline 100mg 1 tab twice daily and Prednisone placebo 1 tab once daily
  Other Names: Prednisone placebo 1 tab once daily in arms 1 and 2
  Arms: Low-dose theophylline arm; Placebo
Drug: Placebo (for Theophylline) — One tablet twice daily in arm 1 (theophylline placebo 1 BD + prednisone placebo 1 once daily)
  Other Names: Theophylline placebo 1 tab twice daily
  Arms: Placebo

SUMMARY:
The aim of this multi-centre, double blind, randomised, controlled trial (DBRCT) is to assess the effect of low dose theophylline, singly and in combination with low dose oral prednisone, on COPD (Chronic Obstructive Pulmonary Disease) exacerbations, quality of life and secondary clinical outcomes compared with usual therapy and placebo over 48 weeks of treatment. 1670 symptomatic patients with COPD will be recruited in China for comparison of low dose theophylline versus placebo and low dose theophylline + low dose prednisone The primary end-point for this study is the annualised COPD exacerbation rate between the treatment groups. Secondary outcomes included time to first severe exacerbation requiring hospitalisation or death, health status, and pre- and post-bronchodilator spirometry.

DETAILED DESCRIPTION:
The investigators hypothesise that patients with COPD will have beneficial responses to low dose theophylline and prednisone, superior to placebo and low dose theophylline alone, reflected by a range of clinical outcomes.

The study aims to demonstrate that treatment with low dose oral prednisone and low dose, slow release theophylline compared to low dose, slow release theophylline only or placebo will reduce COPD exacerbations and improve a range of secondary outcomes including quality of life, COPD Assessment Test (CAT) score, hospital admissions and lung function.

Eligible participants will be randomised to one of three treatment arms in a DBRCT and will receive placebo OR low-dose theophylline (100 mg twice a day) OR low-dose theophylline 100 mg twice a day (BD) plus low-dose prednisone (5 mg once a day)

Patients will be eligible for inclusion if all the following criteria are met:

* Current or former smokers (>10 pack years) or biomass exposure
* 40 - 80 years of age
* Clinical diagnosis of COPD
* Post-bronchodilator forced expiratory volume at one second (FEV1) <70% predicted
* Post bronchodilator FEV1/forced vital capacity (FVC) ratio<0.7

ELIGIBILITY:
Inclusion Criteria:

* Current or former smokers (> 10 pack years) or biomass exposure
* 40 - 80 years of age
* Clinical diagnosis of COPD
* Post-bronchodilator FEV1 < 70% predicted
* Post bronchodilator FEV1/FVC ratio < 0.7

Exclusion Criteria:

* Life expectancy of less than 12 months
* Exacerbation or respiratory infection within 4 weeks prior to randomisation
* Patient is taking and requires maintenance oral corticosteroids
* Patient is on domiciliary oxygen
* There has been previous pulmonary resection
* Previous sensitivity to, or intolerance of theophylline
* Coexistent illness precluding participation in the study (epilepsy, chronic liver disease, unstable cardiovascular disease, diabetes, active malignancy)
* Inability to complete quality of life questionnaire
* Concomitant major illness that would interfere with visits, assessments and follow-up
* Have evidence of chronic liver disease, or transaminase or gamma-glutamyltransferase (GGT) elevation > 1.5 x upper limit of normal (ULN)
* Random blood glucose level > 8mmol/L
* High chance in the view of the treating physician that the patient will not adhere to study treatment and follow up

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1670 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2018-05-14 (Actual); Study Completion 2018-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Berend, MD, Principal Investigator — The George Institute; Christine R Jenkins, MD, Principal Investigator — The George Institute
Locations (1):
- The George Institute for Global Health, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jenkins CR, Wen FQ, Martin A, Barnes PJ, Celli B, Zhong NS, Zheng JP, Scaria A, Di Tanna GL, Bradbury T, Berend N; TASCS study investigators. The effect of low-dose corticosteroids and theophylline on the risk of acute exacerbations of COPD: the TASCS randomised controlled trial. Eur Respir J. 2021 Jun 10;57(6):2003338. doi: 10.1183/13993003.03338-2020. Print 2021 Jun. PMID 33334939

RESULTS

PARTICIPANT FLOW:
Groups:
- Low-dose Theophylline Arm: Theophylline 100 mg twice daily
  Theophylline: Theophylline is an oral methylxanthine which relaxes smooth muscle through its action as a phosphodiesterase inhibitor
  Placebo (for prednisone): - Arm 1 : Theophylline Placebo 1 tab twice daily and Prednisone placebo 1 tab once daily
  - Arm 2 : Theophylline 100mg 1 tab twice daily and Prednisone placebo 1 tab once daily
- Placebo: Placebo theophylline, one tablet twice daily, and Placebo prednisone, one tablet once daily
  Placebo (for prednisone): - Arm 1 : Theophylline Placebo 1 tab twice daily and Prednisone placebo 1 tab once daily
  - Arm 2 : Theophylline 100mg 1 tab twice daily and Prednisone placebo 1 tab once daily
  Placebo (for Theophylline): One tablet twice daily in arm 1 (theophylline placebo 1 twice daily + prednisone placebo 1 once daily)
Period: Overall Study
Arm/Group | Low-dose Theophylline Arm | Placebo | Theophylline and Prednisone Arm
Started | 568 | 554 | 548
Completed | 411 | 408 | 423
Not Completed | 157 | 146 | 125

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo theophylline, one tablet twice daily, and Placebo prednisone, one tablet once daily
  Placebo (for prednisone): - Arm 1 : Theophylline Placebo 1 tab twice daily and Prednisone placebo 1 tab once daily
  - Arm 2 : Theophylline 100mg 1 tab twice daily and Prednisone placebo 1 tab once daily
  Placebo (for Theophylline): One tablet twice daily in arm 1 (theophylline placebo 1 BD + prednisone placebo 1 once daily)
- Total: Total of all reporting groups
Arm/Group | Placebo | Low-dose Theophylline Arm | Theophylline and Prednisone Arm | Total
Number analyzed (Participants) | 554 | 568 | 548 | 1670
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (8.5) | 64.4 (7.8) | 64.9 (7.7) | 64.4 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 134 | 144 | 406
  Male | 426 | 434 | 404 | 1264
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 554 | 568 | 548 | 1670
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 554 | 568 | 548 | 1670
Current Smoker [Count of Participants; unit: Participants] | 98 | 121 | 113 | 332
Pack Years - Current Smoker [Mean (Standard Deviation); unit: years] | 43.5 (27.1) | 40.5 (22.3) | 44.4 (22.7) | 42.7 (23.9)
Spirometry - Pre bronchodilator Forced Expiratory Volume in one second (FEV1) [Mean (Standard Deviation); unit: L/sec] | 1.0 (0.4) | 1.0 (0.4) | 0.9 (0.4) | 1.0 (0.4)

OUTCOME MEASURES:

1. Primary Outcome: Total COPD Exacerbation Rate
Description: The total number of COPD exacerbations reported within 48 weeks
Time Frame: 48 weeks observation; rate annualised
Measure: Number (95% Confidence Interval); unit: Exacerbations per participant year
Arm/Group | Placebo | Low-dose Theophylline Arm | Theophylline and Prednisone Arm
Number analyzed (Participants) | 554 | 568 | 548
Exacerbations per participant year | 1.00 [0.87 to 1.14] | 0.86 [0.75 to 0.99] | 0.89 [0.78 to 1.02]

2. Secondary Outcome: Time to First COPD Exacerbation
Description: The median time (days) from randomisation to first exacerbation per participant
Time Frame: Median time (days) from randomisation to first exacerbation over a 48 week period per participant
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo | Low-dose Theophylline Arm | Theophylline and Prednisone Arm
Number analyzed (Participants) | 554 | 568 | 548
Days | 137 [58.5 to 233.5] | 150 [66.0 to 242.0] | 151 [71.0 to 247.0]

3. Secondary Outcome: Quality of Life Measured by St. George's Respiratory Questionnaire (SGRQ)
Description: THe St. George's Respiratory Questionnaire (SGRQ) is a disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease. Scores range from 0 to 100, with higher scores indicating more limitations.
Time Frame: Change over 48 week study duration
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Low-dose Theophylline Arm | Theophylline and Prednisone Arm
Number analyzed (Participants) | 554 | 568 | 548
Scores on a scale | -4.95 (0.91) | -6.85 (0.91) | -6.48 (0.89)

4. Secondary Outcome: Post Bronchodilator FEV1
Description: The change in post bronchodilator FEV1 from baseline to 48 weeks
Time Frame: Change at 48 weeks
Measure: Mean (Standard Deviation); unit: L/sec
Arm/Group | Placebo | Low-dose Theophylline Arm | Theophylline and Prednisone Arm
Number analyzed (Participants) | 554 | 568 | 548
L/sec | -0.02 (0.01) | -0.01 (0.01) | -0.02 (0.01)

5. Secondary Outcome: Change in COPD Assessment Test (CAT) Score
Description: The COPD Assessment Test (CAT) is a patient-completed questionnaire assessing globally the impact of COPD (cough, sputum, dysnea, chest tighteness) on health status. The range of CAT scores from 0-40. Higher scores denote a more severe impact of COPD on a patient's life. The outcome measure is assessing the change in score from baseline to 48 weeks. A negative change denotes an improvement in health status.
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Low-dose Theophylline Arm | Theophylline and Prednisone Arm
Number analyzed (Participants) | 554 | 568 | 548
Score on a scale | -2.29 (0.33) | -2.77 (0.33) | -2.57 (0.33)

6. Other Pre Specified Outcome: Hospitalisations
Description: The total number of hospitalisation events within 48 weeks
Time Frame: 48 weeks
Measure: Number; unit: Number of hospitalisation events
Arm/Group | Placebo | Low-dose Theophylline Arm | Theophylline and Prednisone Arm
Number analyzed (Participants) | 554 | 568 | 548
Number of hospitalisation events | 120 | 101 | 122

ADVERSE EVENTS:
Time Frame: Adverse events were collected from all participants over the 48 weeks of the intervention period.
Arm/Group | Placebo | Low-dose Theophylline Arm | Theophylline and Prednisone Arm
All-Cause Mortality (participants affected / at risk) | 3/554 | 2/568 | 2/548
Serious Adverse Events (participants affected / at risk) | 96/554 | 91/568 | 83/548
Other Adverse Events (participants affected / at risk) | 196/554 | 222/568 | 202/548
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=554) | Low-dose Theophylline Arm (N=568) | Theophylline and Prednisone Arm (N=548)
COPD Exacerbation - Hospitalised (Respiratory, thoracic and mediastinal disorders) | 96 (135) | 91 (102) | 83 (115)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=554) | Low-dose Theophylline Arm (N=568) | Theophylline and Prednisone Arm (N=548)
COPD Exacerbation - not hospitalised (Respiratory, thoracic and mediastinal disorders) | 168 (306) | 181 (290) | 173 (306)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 28 (37) | 41 (54) | 29 (34)

LIMITATIONS AND CAVEATS:
There are some limitations to our study, there was a 26% withdrawal rate in this study, with a higher rate of withdrawals occurring earlier in the trial. Patients requested withdrawal if they felt the treatment was not helping them and, in particular, if they suffered an exacerbation. This was most evident at the first study visit after treatment commencement, when the greatest number of withdrawals occurred.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All papers will be authored by all or a subgroup of members of the TASCS Publications Committee. Publications prior to the primary and major secondary papers may only be initiated by the Publications Committee. Publications subsequent to the primary and major secondary papers may be authored by individually named authors, and may at the request of the Publication Committee be required to include the annotation "On behalf of the Theophylline and Steroids in COPD (TASCS) trial investigators".

DOCUMENTS (2):
  • Study Protocol (2015-05-27): https://cdn.clinicaltrials.gov/large-docs/27/NCT02261727/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/27/NCT02261727/SAP_001.pdf